CLINICAL TRIAL: NCT04400110
Title: Shortened Antibiotic Therapy for Febrile Urinary Tract Infection (UTI) in Childhood: a Multicenter Randomized Controlled Trial
Brief Title: Short Therapy for Febrile UTI in Childhood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC 10/18
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infections
Keywords: short antibiotic therapy; urinary tract infection; children
MeSH Terms: conditions — Urinary Tract Infections | interventions — Amoxicillin; Clavulanic Acid; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short treatment group (Experimental): Amoxicillin and clavulanic acid 50 mg/kg three times daily administered orally for 5 consecutive days
  Interventions: Drug: Amoxicillin and Clavulanic Acid in Oral Dose Form
- Standard treatment group (Active Comparator): amoxicillin and clavulanic acid 50 mg/kg three times daily administered orally for 10 consecutive days
  Interventions: Drug: Amoxicillin and Clavulanic Acid in Oral Dose Form

INTERVENTIONS:
Drug: Amoxicillin and Clavulanic Acid in Oral Dose Form — 50 mg/kg three times daily administered orally

SUMMARY:
Febrile urinary tract infections (UTIs) are common in children, but there is no consensus concerning the duration of the antibiotic treatment. Current recommendations include the use of an oral antibiotic, chosen between amoxicillin and clavulanic acid or a third-generation cephalosporin (ceftibuten), for a minimum of seven to a maximum of 14 days. In an antibiotic overuse-sparing model, proper evaluation of a shorter therapy in the treatment of febrile UTI in childhood is lacking.

The objective of this randomized controlled trial is to assess the non inferiority of a five days oral course of amoxicillin and clavulanic acid vs the standard 10-day regimen in the treatment of febrile UTIs in children.

The trial results might provide evidence of the non-inferiority of a short duration of the antibiotic course for the treatment of febrile UTI in childhood, contributing to a reduction in the over-use of antibiotics and consequently limiting the emergence of antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 3 months to 5 years;
2. Clinical diagnosis of febrile UTI, defined by fever ≥38°C and positive result of urinalysis (nitrite and/or leukocyte esterase positivity) in two consecutive urine samples collected by bladder catheterization or clean catch (19). The diagnosis of UTI will be then confirmed by positive urine culture for a single type of bacterium with a charge> 105 CFU /ml as per the Recommendations of the Italian Society of Pediatric Nephrology (SINePe) (19).

Exclusion Criteria:

1. "Complicated" febrile UTI (septic appearance, repeated vomiting impeding oral administration of the antibiotic, severe-moderate dehydration with the need for intravenous antibiotic therapy)
2. Presence of an inserted urinary catheter
3. Immunodeficiency
4. Hypersensitivity to the active substance or other beta-lactam antibiotics
5. Any antibiotic treatment received in the previous 15 days.
6. Presence of another poorly controlled chronic medical condition (diabetes, inflammatory bowel disease, etc.)
7. Presence of neurological bladder
8. Presence of phenylketonuria or glucose-galactose malabsorption
9. Intestinal malabsorption
10. Poor compliance
11. History of jaundice or liver failure positive

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of infection recurrence | within 30 days after the end of the intervention
  Infection recurrence rate is defined as the reappearance of signs and symptoms of febrile UTI by the first day after the end of antibiotic therapy

SECONDARY OUTCOMES:
Rate of complete resolution of signs and symptoms | within 30 days after the end of the intervention
  The complete resolution of the signs and symptoms (clinical assessment and urinalysis) related to the infection evaluated at the end of the treatment, without the need for additional or alternative antibiotic therapy (short term clinical efficacy)
Rate of antibiotic-resistant or of opportunistic strains in relapses | within 30 days after the end of the intervention
  Antibiotic resistance is defined as the presence of positive urinalysis and positive urine culture for a single type of bacterium resistant to amoxicillin and clavulanic acid, after treatment in case of relapse. The bacterial growth will be considered significant if >105 colony-forming unit/ml (CFU/ml) (>104 CFU/ml for urine samples collected by bladder catheterization). Urine cultures containing more than one bacterial species will be considered contaminated.

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD Prof, Study Chair — Institute for maternal and child health Burlo Garofolo; Marco Pennesi, MD, Principal Investigator — Institute for maternal and child health Burlo Garofolo
Locations (13):
- Italy (13):
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Santa Maria delle Croci Hospital, Ravenna, Emilia-Romagna
  - Ospedale San Polo, Monfalcone, Friuli Venezia Giulia
  - Pediatric Department, Santa Maria degli Angeli Hospital, Pordenone, Friuli Venezia Giulia
  - Institute for Maternal and Child Health IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia
  - ASUIUD Azienda sanitaria universitaria integrata di Udine, Udine, Friuli Venezia Giulia
  - Fondazione Policlinico Agostino Gemelli - IRCCS City Rome, Rome, Lazio
  - Fondazione IRCSS Ca Granda, Policlinico di Milano, Milan, Lombardy
  - A.O.U.G. Martino, Messina, Sicily
  - Ospedali Riuniti di Ancona - Ospedale Salesi, Ancona, The Marches
  - San Martino Hospital, Belluno, Veneto
  - Department of Woman and Child Health, University of Padua City, Padua, Veneto
  - UOC Pediatria Ospedale Ca' Foncello, Treviso, Veneto

IPD SHARING:
Plan to Share IPD: No